CLINICAL TRIAL: NCT05116371
Title: Control of Bleeding on Nexplanon in Latinx Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Holly Bullock, Assistant Professor, Department of OBGYN, University of Arizona
Other Study IDs: IRB 2104687928
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Contraception
Keywords: etonogestrel implant; irregular bleeding
MeSH Terms: interventions — Contraceptives, Oral, Combined

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Same day initiation option: 1) ENG implant with initiation of concurrent COC use for bleeding control at time of insertion
  Interventions: Drug: 150 mcg levonorgestrel/30 mcg ethinyl estradiol
- Group 2: Delayed initiation option: 2) ENG implant alone with option for "delayed initiation" of COC if bleeding concerns develop
  Interventions: Drug: 150 mcg levonorgestrel/30 mcg ethinyl estradiol

INTERVENTIONS:
Drug: 150 mcg levonorgestrel/30 mcg ethinyl estradiol — concurrent use of COC with Nexplanon
  Other Names: combined oral contraceptive (COC)

SUMMARY:
In this study, researchers want to find out more about how the Etonogestrel (ENG) contraceptive implant device (also known as Nexplanon) changes people's periods. Study subjects will self select into an exposure group- starting combined hormonal contraceptive pills (COC) on the same day as Nexplanon placement or a "delayed initiation" of COC when/if bleeding concerns develop. Patients will be followed for 12 months.

DETAILED DESCRIPTION:
The study will be conducted at University of Arizona. Investigators will recruit people seeking Nexplanon placement and willing to enroll. We aim to enroll 144 patients.

Visit 1:

All patients ages 14-24 presenting for contraception services will be screened for potential inclusion. A trained research assistant will conduct a brief patient-centered contraceptive counseling session focusing on patient preferences.

If interested in participating, the patient will be given a card to present to their clinician. During the visit, patient and provider will discuss further method selection including risks, benefits, and alternatives. The clinician will assess for contraindications per the CDC MEC for use of COC or the implant. Screening for pregnancy, sexually transmitted infections, and cervical cancer screening will follow as clinically indicated. If pregnancy test is negative and clinician can be reasonably certain that patient is not pregnant using the CDC Selected Practice Recommendations, the ENG implant will be placed.

After a clinician encounter, the research assistant will consent those interested in participating. Patients will be assigned a unique identification number once they self-select into their exposure group of choice:

1. ENG implant with initiation of concurrent COC use for bleeding control at time of insertion
2. ENG implant alone with option for "delayed initiation" of COC if bleeding concerns develop

Enrolled patients will complete Demographic Questionnaire and Bleeding Preference Questionnaire.

Enrolled patients in exposure group 1 will receive 6 months COC pills (150 mcg levonorgestrel/30 mcg ethinyl estradiol) and condoms for the first week of back-up method. After 6 months, they will be offered a prescription to continue COC pills. Patients in exposure group 2 will be receive handouts describing how to contact the research team should bleeding concerns develop. A telehealth or in-person visit will be arranged with the research clinicians, during which the patient may opt to start COC pills. A 6 month supply will be provided.

Follow-Up:

Follow-up contact will be weekly for the first 6 months. There will also be 9 and 12 month contact.

Each contact will be a brief text-message survey inquiring about bleeding patterns, pill usage and side effects. The ENG implant will be removed upon request at any time during the study.

Study participation will be completed after the 12 month follow-up survey.

No blood draws will occur during this study.

There is little data available on the adverse effects of ENG implant use and combined COC. This is a common clinical practice to combine use for bothersome bleeding and this study will collect long-term data regarding this practice.

ELIGIBILITY:
Inclusion Criteria:

Fluent in English or Spanish Access to a cellular phone with text messaging and internet capabilities Capable of and willing to receive cellular phone text message Interest in preventing pregnancy for at least 12 months with the ENG implant Interest in use of COC pills with concurrent with ENG implant use Negative urine pregnancy test

Exclusion Criteria:

Contraindication to COC pills or ENG implant as determined by the Centers for Disease Control Medical Eligibility Criteria for Contraceptive Use (CDC MEC) Less than 4 weeks postpartum

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: University of Arizona is a federally designated Hispanic Serving Institution with 28% of its undergraduate population self-identifying as Hispanic. The Department of Obstetrics and Gynecology provides a large proportion of contraceptive care in southern Arizona and is situated to serve as an incubator for participatory research with our Latinx community. From 7/1/2018 - 7/1/2019, a total of 340 patients had implants placed, with 50% of those patients identifying as Latinx or Hispanic. Over a 24 months enrollment period, we estimate that approximately 600 people will want an ENG implant, and through screening that 50% will meet inclusion criteria (300), and 50% will consent to participate (150). Our target for enrollment in 144 (72 non-Latinx and 72 Latinx).
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
bleeding pattern preferences (measurement: questionnaire) | 12 months
  Evaluate the bleeding pattern preferences of people prior to contraception initiation

SECONDARY OUTCOMES:
acceptability (measurement: questionnaire and follow-up surveys) | 12 months
  willingness to initiate concurrent use of COC pills with ENG implant
continuation (measurement: follow-up surveys) | 12 months
  duration of concurrent use of COC pills with ENG implant; continuation of implant
bleeding patterns (measurement: follow-up surveys) | 12 months
  bleeding patterns with concurrent use of COC pills with ENG implant
side effects (measurement: follow-up surveys) | 12 months
  side effects with concurrent use of COC pills with ENG implant

IPD SHARING:
Plan to Share IPD: No